CLINICAL TRIAL: NCT01174277
Title: Immunological Changes in Chronic Graft Versus Host Disease Treated With Extracorporeal Photopheresis
Brief Title: Pilot Study: Patients With Chronic Active Graft Versus Host Disease That Have Failed or Not Tolerated Standard Therapy.
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12179
Record Dates: First submitted 2010-07-27; First posted 2010-08-03 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Blood Stem Cell Transplant Failure; Graft Versus Host Disease
Keywords: chronic graft versus host disease; transplant; stem cell
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected at study entry and at 2, 4, 6 and 12 months following treatment
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Collection of blood sample: Blood draw
  Interventions: Other: Collection of blood sample

INTERVENTIONS:
Other: Collection of blood sample — Participation involves collection of blood sample at baseline, 2, 4, 6 and 12 months regardless of whether or not patients continue on treatment.

SUMMARY:
By doing this study, researchers hope to understand the many changes that occur in the blood of people who have chronic GvHD. This may also help the researcher understand how ECP works and help guide therapy for patients who have chronic GvHD in the future.

DETAILED DESCRIPTION:
The occurrence of acute or chronic graft-versus-host disease (GVHD) and its prevention/treatment induce further immunologic compromise. Graft-versus-host disease (GvHD) accounts for significant morbidity and mortality in recipients of allogeneic bone marrow transplants (BMT) or peripheral blood stem cell (PBSC) transplants. The condition occurs as donor lymphocytes recognize the recipient's tissue as foreign and mount an inflammatory and destructive response in the recipient. GvHD has a predilection for epithelial tissues, especially skin, liver, and the mucosa of the gastrointestinal tract. This can lead to severe skin lesions, gastrointestinal hemorrhage, and liver failure. In addition, people with GvHD are especially susceptible to infection. Approximately 30-70% of people undergoing allogeneic HSCT for hematologic malignancies can anticipate experiencing acute and/or chronic GVHD. The physical consequences depend on the severity of GVHD, but moderate to severe organ system involvement is associated with substantial medical morbidity and mortality. The current standard of care treatment for patients with chronic graft-vs-host disease is steroid treatment with or without a calcineurin inhibitor. This treatment, while effective for some, does not control the chronic gvhd of all. The use of extracorporeal photopheresis (ECP) was developed in patients with several inflammatory and autoimmune diseases, including scleroderma and rheumatoid arthritis. Successful use of ECP has also been reported in patients with cutaneous T cell lymphoma, the Sezary syndrome variant, cardiac and lung transplant rejection and other T cell mediated/autoimmune and autoimmune diseases and even after facial transplantation. More recently, ECP has proven to be a highly effective useful tool in the treatment of GvHD.

The exact mechanism of action of ECP is unknown, but the principle of the process is to induce leucocyte apoptosis with UVA radiation after their exposure to psoralens, which are light sensitizers. These leukocytes are immediately re-infused into the patient, where they undergo early apoptosis. Following apoptosis, the leukocytes are engulfed by macrophage or other antigen-presenting cells, such as immature dendritic cells, in an anti-inflammatory cytokine environment. The anti-inflammatory cytokine secretion pattern, with a switch from TH1 to TH2 for CD4+ lymphocytes, and the engulfment by immature cells without co-stimulatory molecules induces anergy, by deleting effector T-cells that responded to the presented antigens. An increase in regulatory T-cells (T-regs) is also induced after ECP and may contribute to allograft acceptance by the recipient.

ECP has also been effective in treating solid organ transplant rejection and improving the course of various autoimmune diseases, such as rheumatoid arthritis, systemic lupus erythematosis, and pemphigus vulgaris. Since the early 1990s, ECP has been investigated as a rescue immunotherapy for patients with steroid resistant acute and chronic GVHD. ECP is generally well tolerated and Phase II data have confirmed activity in more than 250 patients with steroid-refractory cGVHD.

ECP involves the isolation of peripheral blood buffy coat cells, ex vivo exposure of the cells to 8-methoxypsoralen (8-MOP) and ultraviolet-A radiation, and subsequent re-infusion of the treated cells to the patient. The combination of 8-MOP and PUVA results in DNA crosslinks and causes apoptosis. However, the direct induction of lymphocyte apoptosis is unlikely to account for the clinical efficacy of ECP given that less than 10% of circulating leukocytes are exposed to PUVA during ECP.

The mechanism of ECP beyond the effects of apoptosis induction is incompletely understood. Studies to date suggest that ECP in autoimmune conditions or GVHD stimulates anti-idiotypic responses against host tissue-reactive T cell clones, attenuates antigen-presenting function by type 2 dendritic cells, and induces anti-inflammatory cytokine responses. In addition, an important component of tolerance induction is thought to involve the expansion of Tregs that suppress alloreactive mechanisms.

ECP therapy has been studied in two well-defined minor MHC incompatible murine models of CD8+ or CD4+ T cell mediated GVHD. These studies showed that ECP treated cells could successfully reverse established GVHD by reducing allogeneic responses of donor effector T cells and generating FOXP3+ Tregs from donor cells that had not been directly exposed to PUVA, thereby ruling out a mechanistic role for direct apoptosis of effector cells. The increase in Tregs occurred early after the infusion of ECP treated cells, remained stable for several weeks, and was required to reduce GVHD and mortality after BMT. Correlative data in humans is preliminary, but one small case series has shown an increase in the percentage of functional Tregs after 6 ECP procedures from 8.9% to 29% of the total circulating CD4+ cells (p = .05). UVAR Photopheresis System (Therakos, Inc., Exton, PA, USA) was approved for ECP treatment of advanced cutaneous T cell lymphoma in 1988 by the Food and Drug Administration. In 2009 FDA approval was granted for this indication for the new Cellex machine.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT recipients who have chronic extensive GvHD and who have failed or have not been able to tolerate conventional therapy
* Platelets ≥ 20,000 without transfusion support
* Weight ≥ 15 kg.
* Stated willingness to use contraception in women of childbearing potential

Exclusion Criteria:

* Patients who may not be able to tolerate ECP
* Patients who have received Rituximab monoclonal antibody therapy in the past 3 months
* Patients with a known hypersensitivity to psoralens
* Pregnant or breastfeeding
* Patients who are unable to sign informed consent or who do not have a representative to give permission to participate

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone allogeneic HSCT and are being managed for chronic Graft versus Host Disease by the University of Kansas Blood and Marrow Transplantation Program, and the Children's Mercy Hospital BMT program, will be invited to take part in the study.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Determine effects of ECP using Cellex on T and B cell subsets and CD4+ cell differentiation | 2 years
  Flow cytometry will be used to characterize T and B cell subsets in the blood of ECP patients. We will also isolate CD4+ T cells from ECP patients, stimulate the cells in culture, and measure proliferation and cytokine production. These assays will be performed prior to ECP therapy and at two, four and six months following ECP therapy.

SECONDARY OUTCOMES:
To correlate the effects of ECP on immunologic parameters with clinical outcomes. | 2 years
  We will measure serum levels of eight biomarkers known to correlate with GvHD and evaluate the patients for clinical signs of GvHD. The biomarkers and clinical signs will be correlated with the immunologic parameters described in the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Abhyankar, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Mercy Hospital, Kansas City, Missouri